CLINICAL TRIAL: NCT05589025
Title: Pulpotomy Versus Pulpectomy in Carious Vital Pulp Exposure of Primary Incisors: Randomized Controlled Trial
Brief Title: Pulpotomy Versus Pulpectomy in Vital Primary Incisors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Research Centre, Egypt (Other)
Collaborators: Cairo University (Other)
Responsible Party: Principal Investigator, Lamia Mohamed Khairy Gadallah, Researcher, National Research Centre, Egypt
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 14154
Record Dates: First submitted 2022-10-10; First posted 2022-10-21 (Actual); Last update posted 2022-10-21 (Actual); Status verified 2022-10

CONDITIONS: Dental Caries; Pulp Disease, Dental
Keywords: pulpotomy; pulpectomy; tooth, deciduous
MeSH Terms: conditions — Dental Caries; Dental Pulp Diseases | interventions — formocresol; Zinc Oxide; Eugenol

STUDY DESIGN:
Intervention Model Description: split mouth
Who Masked: Participant, Outcomes Assessor
Masking Description: blinding of assessor of clinical outcomes
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- treatment group (Active Comparator): pulpotomy: amputation of coronal pulp
  Interventions: Procedure: pulpotomy technique with formocresol
- control group (Active Comparator): Pulpectomy: complete removal of the pulp tissues from the canals
  Interventions: Procedure: pulpectomy technique with zinc oxide and eugenol

INTERVENTIONS:
Procedure: pulpotomy technique with formocresol — The pulpotomy procedure performed was a modification of that described by Pinkham et al; 2005 where pulp chamber was unroofed using a no. 330 sterile bur in a water-cooled high-speed handpiece. The entire roof of pulp chamber and overhanging dentinal remnants over the pulp horns were removed. After the completion of the access cavity, coronal pulp was extirpated using a sharp excavator. Any residual coronal pulpal tissue was removed using a sterile round bur in a slow-speed handpiece to a depth of few millimeters below the free gingival margin. Hemostasis was achieved with a water-dampened cotton pellet. If hemostasis was not achieved after the initial application of the cotton pellet, the case was eliminated from the study. Following hemostasis, a cotton pellet, moistened with formocresol was applied for 3 minutes and removed. A zinc- oxide and eugenol base was placed over the amputation site. Thereafter, a glass ionomer base was applied.
  Other Names: vital pulp therapy
  Arms: treatment group
Procedure: pulpectomy technique with zinc oxide and eugenol — The pulpectomy procedure used herein was a modification of that described by Payne et al;1993 Pulp chamber was unroofed using a no. 330 sterile bur in a water-cooled high-speed handpiece. The entire roof of pulp chamber and overhanging dentinal remnants over the pulp horns were removed. An initial endodontic K-file fitting snugly in the canal was introduced inside it. In most cases, the pulp tissue was removed completely on the first attempt. If the first attempt was unsuccessful, the procedure was repeated and canals were generally enlarged three sizes past the initial file to eliminate the organic remnants. Copious irrigation with a light flow of sterile 0.9% NaCl-solution was used throughout the procedure. At the end, the canals were dried and filled with zinc-oxide & eugenol.
  Other Names: root canal treatment
  Arms: control group

SUMMARY:
The aim of this split mouth randomized controlled study was to compare formocresol pulpotomy and zinc-oxide and eugenol pulpectomy in the treatment of vital pulp exposure in primary incisor. 39 Contralateral pairs of incisors were randomly assigned to receive pulpotomy or pulpectomy in children aged from 18 to 66 months old.

Clinical and radiographical evaluations were performed at 6 and 12 months

DETAILED DESCRIPTION:
* This randomized controlled trial with split mouth design
* The study was approved by the research ethics committee of the National research centre.
* Participants in this study were recruited from August 2015 till December 2016. Patients' eligibility criteria were medically free patients, aging from 18 to 66 months old, with two or more carious vital primary maxillary incisors where exposure of the vital pulp following the removal of dental caries was inevitable.
* Sample size was calculated using PS Computer Program .A study of matched cases and controls was planned. Prior data indicated that success rates among controls were 0.78 . If the true success rate for experimental subjects is 1, then we needed to study 31 pairs to be able to reject the null hypothesis that the success rates for experimental and control subjects are equal with probability (power) 0.8. The Type I error probability associated with this test of this null hypothesis is 0.05.McNemar's chi-squared statistic was used to evaluate this null hypothesis. This number has been increased to a total sample size 39 in each group, to allow for losses of around 25%.
* The procedure, possible discomforts or risks, as well as possible benefits were explained completely to the parents or legal guardians, and they were allowed to sign in the patients' ethics form.
* The child participants and legal guardian of each participating child were blinded to the type of treatment they received while it was not possible for the operator or the radiographic assessors to be blinded due to the nature of the treatment received.
* An incisor in each pair was randomly assigned by a coin toss to either the intervention (pulpotomy group) on the head side or the control (pulpectomy group) on the tail side with the contralateral paired incisor being designated to the other treatment group.
* Clinical examination and preoperative periapical radiographs were performed for eligible patients. After induction of anesthesia, teeth were properly isolated with cotton rolls and suction as rubber dam was not tolerated by children less than 6 years of age. Complete removal of caries or undermined enamel was performed before access cavity preparation.•
* For follow up: Clinical evaluation was performed on all primary incisors during the follow-up visits at one, six and twelve months post-operatively while radiographic evaluation was performed at six and twelve months follow up visits
* For radiographic evaluation, the radiographs were taken with a size 0 or 1 periapical films (D-speed Film, Ultra-speed Carestream Dental,USA) using the bisecting angle technique. The radiographs were scanned on a viewer and transmitted to a computer hardware to be properly saved. The evaluation was performed by two independent assessors and differences were solved by consensus. Data analysis was performed on the consensus scores.
* For Statistical analysis, Chi square test was used to compare between the two groups. The significance level was set at P ≤ 0.05. Also estimated effect size was calculated with 95% Confidence Interval. Kaplan-Meier used for survival analysis. Statistical analysis was performed with IBM® SPSS® (SPSS Inc., IBM Corporation, NY, USA) .

ELIGIBILITY:
Inclusion Criteria:

* Two or more carious vital primary maxillary incisors where exposure of the vital pulp following the removal of dental caries was inevitable.
* No history of spontaneous pain
* No lingering provoked pain
* No pain on percussion, No fistula, or sinus tract
* No history of trauma
* No periapical radiolucency
* No pathologic root resorption
* No pulp calcification.

Exclusion Criteria:

* Teeth with physiologic resorption exceeding one-third of the root
* Teeth non-restorable with crowns.

Ages: 18 Months to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 39 (Actual)
Dates: Start 2015-08-01 (Actual); Primary Completion 2016-12-01 (Actual); Study Completion 2016-12-15 (Actual)

PRIMARY OUTCOMES:
clinical failure | 1 year
  composite outcome including pain, soft tissue pathology, and tooth mobility. All are binary outcomes. The presence of any item is recorded as a clinical failure.
radiographic failure | 1 year
  a composite outcome including pathologic mobility and pathologic root resorption. Both are binry outcomes, the presence of any of them is recorded as a radiographic failure.

SECONDARY OUTCOMES:
survival rate | 1 year
  the survival of the tooth in the oral cavity

CONTACTS AND LOCATIONS:
Overall Officials: Lamia Gadallah, Researcher, Principal Investigator — National Research Centre, Egypt

IPD SHARING:
Plan to Share IPD: No
the required data will be published in the study

REFERENCES:
- [Background] Howley B, Seale NS, McWhorter AG, Kerins C, Boozer KB, Lindsey D. Pulpotomy versus pulpectomy for carious vital primary incisors: randomized controlled trial. Pediatr Dent. 2012 Sep-Oct;34(5):112-9. PMID 23211895
- [Background] Aminabadi NA, Farahani RM, Gajan EB. A clinical study of formocresol pulpotomy versus root canal therapy of vital primary incisors. J Clin Pediatr Dent. 2008 Spring;32(3):211-4. doi: 10.17796/jcpd.32.3.ghk26v4554790074. PMID 18524271
- [Background] Smail-Faugeron V, Fron Chabouis H, Durieux P, Attal JP, Muller-Bolla M, Courson F. Development of a core set of outcomes for randomized controlled trials with multiple outcomes--example of pulp treatments of primary teeth for extensive decay in children. PLoS One. 2013;8(1):e51908. doi: 10.1371/journal.pone.0051908. Epub 2013 Jan 3. PMID 23300955
- [Derived] Gadallah LK, Elbardissy A, Elyazeed MA, Alsamad AA, Hamdy M. Pulpotomy versus pulpectomy in carious vital pulp exposure in primary incisors: a randomized controlled trial. BMC Oral Health. 2024 Mar 20;24(1):354. doi: 10.1186/s12903-024-04116-w. PMID 38504243